CLINICAL TRIAL: NCT03648658
Title: Pharmacokinetics and Safety of Treatment With Paracetamol in Children and Adults With Spinal Muscular Atrophy and Cerebral Palsy
Brief Title: Paracetamol Study in Patients With Low Muscle Mass
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mette Cathrine Oerngreen (Other)
Collaborators: Elsass Foundation (Other)
Responsible Party: Sponsor-Investigator, Mette Cathrine Oerngreen, Principal Investigator, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 08-06-2018-paracet; 2018-002295-40 (EudraCT Number)
Record Dates: First submitted 2018-08-08; First posted 2018-08-27 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: SMA II; Cerebral Palsy
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood; Cerebral Palsy | interventions — Acetaminophen; Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Paracetamol 15mg/kg (Experimental)
  Interventions: Drug: Paracetamol 120Mg/5mL Oral Suspension

INTERVENTIONS:
Drug: Paracetamol 120Mg/5mL Oral Suspension — The subjects will be treated with paracetamol in therapeutic doses, 15mg/kg/dose every six hour, with a maximum dosage of 1 g x 4 per day, for three consecutive days.

SUMMARY:
To investigate the safety and toxicity related to paracetamol treatment in children and adults with respectively SMA and CP.

DETAILED DESCRIPTION:
1. Aim

   1. Objectives

      Primary objective:

      The aim of the project is to study the pharmacokinetics of therapeutic doses of paracetamol with specific emphasis on the contributions of the metabolites (glucuronide, sulphate, cysteine and mercapturate), in patients with spinal muscular atrophy(SMA), patients with cerebral palsy(CP), and patients with SMA or CP admitted to the intensive care unit (ICU), in comparison with healthy controls.

      Secondary objective:

      The secondary aim is to compare the safety of paracetamol in patients with SMA, CP and patients with SMA or CP admitted to the ICU, with healthy controls. The investigators would like to assess the influence of age and physiologic covariates (body weight and inflammation markers) on paracetamol pharmacokinetics.
   2. Background Today there are approximately 15.000 patients with neuromuscular disorders in Denmark. This includes the group of patients with muscular wasting. SMA is an example of a neuromuscular disease, where the patients have low skeletal muscle mass. The disease is located in the anterior cells in the spinal cord. This affects the cells that are supposed to send signals about muscle contraction through the nerve pathways, and causes muscle wasting. Spinal muscular atrophy is a hereditary disease caused by a mutation in the Survival Motor Neuron (SMN) 1-gene. SMN is necessary for normal nerve function in the muscles. The patients with SMA have a back-up gene called Survival Motor Neuron (SMN) 2-gene. However, most of the SMN 2-gene cannot be used, because of a missing part in the gene called exon 7. Spinal muscular atrophy is divided into three different types, based on the child's motor skills and when the first symptoms appear. Children with SMA type I experience symptoms within the first six months of life. The children will never experience to sit by themselves without help. They seldom get older than two years; even though it depends on how much intensive respiratory care they receive. The onset of symptoms for children with SMA type II is between 5 and 12 months of age. They usually get diagnosed before they reach the age of 1-2 years. The children will be able to sit by themselves, but will not be able to walk and stand without help. Children with SMA II can get a normal life span. SMA type III is the mildest form. The onset of the symptoms appears after the child is 18 months of age, and the child will be able to walk independently. (1) Cerebral palsy (CP) is another example of a patient group with low muscle weight. CP is caused by a brain damage which occurs either during foetal life, during birth or in the neonatal period. The brain damage occurs in connection to premature birth, oxygen deficiency, infections or blood clots. However, often the specific cause cannot be detected. Every year 180 children with CP are born in Denmark. The disease will not worsen with time, but the symptoms will change gradually as the child grows up. Incorrect positions of joints and bones may occur with time.(2) The investigators have experienced that two patients with SMA II developed acute liver failure, most likely due to paracetamol toxicity. In line with this a case study from 2011 reported that patients with myopathies and muscular atrophies might be at increased risk of toxicity, resulting in acute liver failure, while receiving the recommended dose of paracetamol.(3) Another two cases with similar stories has been described in boys with Duchenne Muscular Dystrophy.(4) Children and young adults with low muscle mass have several risk factors that may increase the susceptibility to paracetamol. First of all, they have a reduced skeletal muscle mass compared to bodyweight.(5) Glutathione (GSH) is a low-molecular-weight thiol, consisting of the amino acids glutamate, cysteine and glycine. Most of the glutathione synthesis occurs in the liver and it is stored in the majority of cells in the body. It has been suggested that skeletal muscle has a remarkable GSH synthesizing ability and high activity of GSH-dependent enzymes. This suggest that skeletal muscle is a major player for the whole body GSH metabolism.(6) We hypothesize that the patients with spinal muscular atrophy, has a lower concentration of glutathione compared to healthy subjects, due to the fact that they have a low skeletal muscle mass. This is relevant because glutathione detoxifies the oxidative metabolite in the paracetamol metabolism. Furthermore, there is a tendency that children and young adults with low muscle mass are malnourished and have a tendency to become critically ill. Several studies have shown that there may be a correlation between malnutrition, fasting, critical illness and glutathione deficiency.(7-9) Lastly, paracetamol is relatively hydrophilic, and the volume of distribution of paracetamol would be further reduced in patients with low muscle mass, thus increasing plasma levels.(10) Paracetamol is commonly used to treat mild-to-moderate pain or to reduce opioid exposure, as part of multimodal analgesia treatment in patients with SMA and CP. In therapeutic doses, about 90% of paracetamol is conjugated in the liver to nontoxic metabolites (glucuronides and sulphates). A small portion (approximately 5 -10 %) is conjugated by cytochrome P450 CYP2E1 to a toxic metabolite, N-acetyl-p-benzo-quinone imin (NAPQI). This metabolite is further conjugated by glutathione to a neutral metabolite and excreted in the urine as cysteine and mercapturate metabolites.(11) In toxic doses, the usual metabolic pathways are overwhelmed; paracetamol is shunted to the cytochrome P450 pathway, and glutathione stores are depleted. Cellular injury and hepatic necrosis occur as NAPQI accumulates.(8) The paracetamol metabolism pathways are slightly different in young children compared to adults. In young children up to 12 years of age, the glucunoride pathway is deficient. The sulphate pathway is the dominant conjugation pathway, and the half-time is prolonged.(12) Patients with low muscle mass may need a lower loading and maintenance doses of paracetamol. However, since only one of the three metabolic pathways of paracetamol (i.e the CYP2E1- mediated pathway) is involved in hepatotoxicity, it is important to explore the separate contributions of the different metabolic pathways.(13) Elevations of alanine aminotransferase (ALT) in the bloodstream are measured as a biomarker, regarding to hepatic events and toxicity. ALT is an enzyme usually found inside the liver cells, however if the liver is damaged or inflamed, it could be released in to the bloodstream. A prospective study of ALT elevations in healthy adults receiving therapeutic doses of paracetamol exists.(14) However, paracetamol kinetics and liver affection has to our knowledge never been studied in patients with low muscle mass before.

   The investigators would like to conduct a prospective study of the safety and toxicity related to paracetamol treatment in children and young adults with respectively SMA and CP.

   This study will provide new and important knowledge about the potential risk involved with paracetamol treatment in therapeutic doses in patients with low muscle mass. If the investigators find that paracetamol in therapeutic doses are toxic in patients with SMA and CP, the results will be implemented in new national and international guidelines for treatment of pain in patients with SMA and CP, to prevent acute liver failure and potential death, thus improving prophylactic care for these patients.
2. Study design

   A prospective, non-randomised, open label, single site clinical trial. Data from the adult patients will be compared to a group of healthy controls for comparison of the primary and secondary outcome measures.

   Data from the children will be compared with data from the literature on healthy children.
3. Study Treatment

The subjects will be treated with paracetamol in therapeutic doses, 15mg/kg/dose every six hour, with a maximum dosage of 1 g x 4 per day, for three consecutive days. Blood samples will be collected before treatment, during the uptake of the first dose, and after the uptake of the first dose of paracetamol. The same procedure will be performed after three days of paracetamol treatment.

ELIGIBILITY:
Inclusion Criteria:

* - Patients: Men, women and children diagnosed with/biochemically verified SMA and CP
* Patients admitted to the ICU: Men, women, children diagnosed with/biochemically verified SMA and CP
* Healthy controls: Need to be healthy, evaluated by the investigator.
* Age:

  * Children: 6-18 years
  * Adult patients: 18-45 years
  * Healthy controls: 18-45 years
  * ICU-admitted patients: 6-45 years
* Signed informed consent to participation in the trial

Exclusion Criteria:

* - Inability to understand the purpose of the trial or cooperate in the conduction of the experiments.

  o For the children this will concern of course the parents or the guardians of the child.
* Competing conditions at risk for compromising the results of the study.
* Participation in other trials that may interfere with the results.
* Intake of medications that may interfere with the results, evaluated by investigator.
* Pregnancy and breastfeeding.
* BMI >30*

  * In morbidly obese patients, the median area under the plasma concentration-time curve from 0 to 8 h. (AUC0-8h) of paracetamol is significantly smaller (p = 0.009), while the AUC0-8h ratios of the glucuronide, sulphate and cysteine metabolites to paracetamol are significantly higher (p = 0.043, 0.004 and 0.010, respectively). In this model, paracetamol CYP2E1-mediated clearance (cysteine and mercapturate) increased with lean body weight.

Ages: 6 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-02-18 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Clearance paracetamol | Three days
  - Clearance (total, glucuronidation, sulphation, CYP2E1 oxidation and unchanged) of paracetamol in patients with SMA, CP and ICU-admitted patients with either SMA or CP
Clearance paracetamol | Three days
  - Clearance (total paracetamol) of paracetamol in patients with SMA, CP and ICU-admitted patients with either SMA or CP
Clearance paracetamol | Three days
  - Clearance (glucuronidation) of paracetamol in patients with SMA, CP and ICU-admitted patients with either SMA or CP
Clearance paracetamol | Three days
  - Clearance (sulphation) of paracetamol in patients with SMA, CP and ICU-admitted patients with either SMA or CP
Clearance paracetamol | Three days
  - Clearance (CYP2E1 oxidation) of paracetamol in patients with SMA, CP and ICU-admitted patients with either SMA or CP
Clearance paracetamol | Three days
  - Clearance (unchanged paracetamol) of paracetamol in patients with SMA, CP and ICU-admitted patients with either SMA or CP
Volume of distribution of paracetamol | Three days
  - Volume of distribution of paracetamol in patients with SMA, CP and ICU-admitted patients with SMA or CP, in comparison with healthy controls.

SECONDARY OUTCOMES:
Liver function tests: ALT, AST, LDH, Alkaline Phosphatase, Bilirubin (U/L) | Three days
  - Liver function tests in patients with SMA, CP and ICU-admitted patients with SMA or CP.: ALT, AST, LDH, Alkaline Phosphatase, Bilirubin (U/L)
Concentration-time data on liver function and paracetamolparametres | Three days
  - Concentration-time data on plasma paracetamol, paracetamol-sulphate, paracetamol-glucuronide, paracetamol-cysteine and paracetamol-mercapturate (oxidative metabolites), plasma-glutathione and liver biomarkers (ALAT, PP, bilirubin, MicroRNA-122 (miR-122)).

CONTACTS AND LOCATIONS:
Overall Officials: Mette Cathrine Ørngreen, MD, DMSc, Principal Investigator — MD
Locations (1):
- Copenhagen Neuromuscular Center, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kolb SJ, Kissel JT. Spinal Muscular Atrophy. Neurol Clin. 2015 Nov;33(4):831-46. doi: 10.1016/j.ncl.2015.07.004. PMID 26515624
- [Background] Rosenbaum P, Paneth N, Leviton A, Goldstein M, Bax M, Damiano D, Dan B, Jacobsson B. A report: the definition and classification of cerebral palsy April 2006. Dev Med Child Neurol Suppl. 2007 Feb;109:8-14. PMID 17370477
- [Background] Ceelie I, James LP, Gijsen V, Mathot RA, Ito S, Tesselaar CD, Tibboel D, Koren G, de Wildt SN. Acute liver failure after recommended doses of acetaminophen in patients with myopathies. Crit Care Med. 2011 Apr;39(4):678-82. doi: 10.1097/CCM.0b013e318206cc8f. PMID 21242792
- [Background] Hynson JL, South M. Childhood hepatotoxicity with paracetamol doses less than 150 mg/kg per day. Med J Aust. 1999 Nov 1;171(9):497. doi: 10.5694/j.1326-5377.1999.tb123758.x. No abstract available. PMID 10615345
- [Background] Orngreen MC, Zacho M, Hebert A, Laub M, Vissing J. Patients with severe muscle wasting are prone to develop hypoglycemia during fasting. Neurology. 2003 Oct 14;61(7):997-1000. doi: 10.1212/01.wnl.0000086813.59722.72. PMID 14557579
- [Background] Sen, C. K. Glutathione: A key role in skeletal muscle metabolism. in Oxidative Stress in Skeletal Muscle 127-139 (Birkhäuser, Basel, 1998). doi:10.1007/978-3-0348-8958-2_8
- [Background] Hammarqvist F, Luo JL, Cotgreave IA, Andersson K, Wernerman J. Skeletal muscle glutathione is depleted in critically ill patients. Crit Care Med. 1997 Jan;25(1):78-84. doi: 10.1097/00003246-199701000-00016. PMID 8989180
- [Background] McClain CJ, Price S, Barve S, Devalarja R, Shedlofsky S. Acetaminophen hepatotoxicity: An update. Curr Gastroenterol Rep. 1999 Feb-Mar;1(1):42-9. doi: 10.1007/s11894-999-0086-3. PMID 10980926
- [Background] Caparrotta TM, Antoine DJ, Dear JW. Are some people at increased risk of paracetamol-induced liver injury? A critical review of the literature. Eur J Clin Pharmacol. 2018 Feb;74(2):147-160. doi: 10.1007/s00228-017-2356-6. Epub 2017 Oct 24. PMID 29067481
- [Background] Pearce B, Grant IS. Acute liver failure following therapeutic paracetamol administration in patients with muscular dystrophies. Anaesthesia. 2008 Jan;63(1):89-91. doi: 10.1111/j.1365-2044.2007.05340.x. PMID 18086077
- [Background] Forrest JA, Clements JA, Prescott LF. Clinical pharmacokinetics of paracetamol. Clin Pharmacokinet. 1982 Mar-Apr;7(2):93-107. doi: 10.2165/00003088-198207020-00001. PMID 7039926
- [Background] Prescott LF. Kinetics and metabolism of paracetamol and phenacetin. Br J Clin Pharmacol. 1980 Oct;10 Suppl 2(Suppl 2):291S-298S. doi: 10.1111/j.1365-2125.1980.tb01812.x. PMID 7002186
- [Background] van Rongen A, Valitalo PAJ, Peeters MYM, Boerma D, Huisman FW, van Ramshorst B, van Dongen EPA, van den Anker JN, Knibbe CAJ. Morbidly Obese Patients Exhibit Increased CYP2E1-Mediated Oxidation of Acetaminophen. Clin Pharmacokinet. 2016 Jul;55(7):833-847. doi: 10.1007/s40262-015-0357-0. PMID 26818482
- [Background] Watkins PB, Kaplowitz N, Slattery JT, Colonese CR, Colucci SV, Stewart PW, Harris SC. Aminotransferase elevations in healthy adults receiving 4 grams of acetaminophen daily: a randomized controlled trial. JAMA. 2006 Jul 5;296(1):87-93. doi: 10.1001/jama.296.1.87. PMID 16820551